CLINICAL TRIAL: NCT03272516
Title: Mindfulness Based Cognitive Therapy (MBCT) for Primary Care Patients With Mild to Moderate Symptoms of Depression or Anxiety.
Brief Title: Mindfulness Based Cognitive Therapy (MBCT) for Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Svala Sigurdardottir, Principal Investigator, University of Iceland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UI-2017-MBCT.
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Depression, Anxiety
Keywords: Mild to moderate Depression; Mild to moderate Anxiety; Mindfulness based cognitive therapy; Primary care; PHQ-9; GAD-7; Antidepressants; Anxiolytica; Subjective wellbeing
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, where patients are randomized to two groups. Group 1 receives treatment as usual, group 2 receives treatment as usual plus Mindfulness Based Cognitive Therapy (MBCT) for symptoms of mild to moderate depression or anxiety.
  Our primary aim is to investigate whether MBCT added to TAU is more effective than TAU alone in reducing mild to moderate symptoms of depression and/or anxiety among primary care patients.
  Our secondary aim is to investigate whether MBCT added to TAU is more effective than TAU alone in:
  1. Increasing subjective wellbeing
  2. Reducing antidepressant/anxiolytica use for primary care patients, with mild to moderate symptoms of depression and/or anxiety.
Who Masked: Investigator
Masking Description: The investigator will contact all participants in both groups via email or telephone to ask them to answer questionnaires.The investigator will not have information about which group which participant is. Participants will be contacted and invited to answer a questionnaire before, after, 6 and 18 months after 8 weeks of TAU and TAU plus MBCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): This group receives treatment as usual (TAU) from his/hers physician. This treatment is different for each physician, but mainly consists of cognitive therapy, personal interviews or antidepressants or anxiolytics.
  Interventions: Other: Treatment as usual (TAU)
- Intervention group (Experimental): Mindfulness Based Cognitive Therapy (MBCT). This group receives 8 weeks of MBCT in addition to usual treatment (TAU). The MBCT consists of weekly group sessions of 2,5 hours, where participants receive cognitive therapy as well as mindfulness meditation. This group is also assigned homework, according to the MBCT protocol..
  Interventions: Behavioral: Mindfulness based cognitive therapy (MBCT); Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Mindfulness based cognitive therapy (MBCT) — Mindfulness Based Cognitive Therapy (MBCT). This group receives 8 weeks of MBCT in addition to usual treatment (TAU). The MBCT consists of weekly group sessions of 2,5 hours, where participants receive cognitive therapy as well as mindfulness meditation. This group is also assigned homework, according to the MBCT protocol.
  Arms: Intervention group
Other: Treatment as usual (TAU) — Usual treatment prescribed by each physician, specifically interview therapy, cognitive therapy, antidepressants and/or anxiolytics as well as a mixture of all of the above.

SUMMARY:
This study is done to evaluate the effects of Mindfulness Based Cognitive Therapy (MBCT) for primary care patients that have mild to moderate symptoms of depression and anxiety. Half of the study participants will receive treatment as usual (TAU), and the other half will receive TAU plus MBCT. The investigators will be comparing changes in symptoms of depression and anxiety between the groups, and hypothesize that the TAU plus MBCT group will have significantly lower symptoms of depression and anxiety compared to TAU group post-intervention

DETAILED DESCRIPTION:
Patients that show mild to moderate symptoms of depression and anxiety are common in the primary care setting. These patients are often treated with antidepressant or anxiolytic medication instead of cognitive therapy, which is the first choice of treatment according to clinical guidelines in Iceland. Although these patients are often referred to cognitive therapy, there are long waiting lists for group therapy and personal therapy is expensive. MBCT has been shown to have good effects on people with recurrent depression and on patients suffering from anxiety. Therefore, the investigators main objective is to assess whether MBCT is effective in the primary care setting for patients with mild symptoms of anxiety and depression and compare its effect to TAU.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 and GAD-7 score 5-14 points
* Age18 - 67
* No current/recent psychotherapy of any kind other than his/hers physicians therapy( can be taking antidepressants but not in CBT)
* No regular meditation or yoga practice
* Not mentally retarded
* Speaks and understands Icelandic
* No current substance dependence
* Not diagnosed with schizophrenic symptoms or bipolar disease that that currently requires treatment
* Not participating in another mental health study

Exclusion Criteria:

1. Age: <18 and >67 years old.
2. Severe psychiatric symptoms requiring psychiatric care
3. Risk of suicide
4. Inability to participate in group sessions because of severe substance misuse;
5. Inability to speak and understand Icelandic
6. Pregnancy;
7. Current psychotherapy of any kind;
8. Participation in any other psychiatric intervention study;
9. Thyroid disease (if newly diagnosed by the doctor).
10. Score under 5 on both GAD7 and PHQ-9 and score over 14 on either GAD7 or PHQ-9.
11. One or more of the following ICD-10 psychiatric diagnoses:

F00-F09 Organic, including symptomatic, mental disorders F10-F19 Mental and behavioural disorders due to psychoactive substance use F20-F29 Schizophrenia, schizotypal and delusional disorders F70-F79 Mental retardation

-

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Symptoms of depression measured with the PHQ-9 questionnaire | up to 18 months
  Comparing scores on the PHQ-9 before and after the intervention as well as, 6 and 18 months after the intervention for both the control group (TAU) and the intervention group (TAU plus MBCT)
Symptoms of anxiety measured with the GAD-7 questionnaire | up to 18 months
  Comparing scores on the GAD-7 before and after the intervention as well as 6 and 18 months after the intervention for both the control group (TAU) and the intervention group (TAU plus MBCT)

SECONDARY OUTCOMES:
Subjective well-being measured with the SWEMWBS questionnaire | up to 18 months
  Comparing overall score on the SWEMWBS before and after the intervention as well as 6 and 18 months after the intervention for both the control group (TAU) and the intervention group (TAU plus MBCT)
Change in use of antidepressants | up to 18 months
  Self reported use of antidepressants in a questionnaire sent out by the study organization
Change in use of anxiolytics | up to 18 months
  Self reported use of antidepressants in a questionnaire sent out by the study organization

CONTACTS AND LOCATIONS:
Overall Officials: Dóra G Gudmundsdóttir, PhD, Study Chair — Directorate of Health, Iceland
Locations (2):
- Iceland (2):
  - Heilsugæslan Grafarvogi, Reykjavik, Grafarvogur
  - Heilsugæslan Miðbæ, Reykjavik

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available to other researchers when requested. We will be willing to share the below mentioned IPD.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and additional data will be shared at the time when the summary data are published or otherwise made available and will be available for 5 years after the end of the study.
Access Criteria: The study protocol, SAP, ICF, CSR and analytic code can be available for relevant researches, working on similar studies or researchers who want to reproduce the protocol and set up of the study as well as for doing a meta-analysis on similar studies. This must be done in the timeframe mentioned above. The group working on this project (the PhD students consult group) will review the requests and make shared decision on that and as well as decide how it will be shared.

REFERENCES:
- [Background] Bados A, Balaguer G, Saldana C. The efficacy of cognitive-behavioral therapy and the problem of drop-out. J Clin Psychol. 2007 Jun;63(6):585-92. doi: 10.1002/jclp.20368. PMID 17457848
- [Background] Stirman SW, Gutierrez-Colina A, Toder K, Esposito G, Barg F, Castro F, Beck AT, Crits-Christoph P. Clinicians' perspectives on cognitive therapy in community mental health settings: implications for training and implementation. Adm Policy Ment Health. 2013 Jul;40(4):274-85. doi: 10.1007/s10488-012-0418-8. PMID 22426739
- [Background] Bondolfi G, Jermann F, der Linden MV, Gex-Fabry M, Bizzini L, Rouget BW, Myers-Arrazola L, Gonzalez C, Segal Z, Aubry JM, Bertschy G. Depression relapse prophylaxis with Mindfulness-Based Cognitive Therapy: replication and extension in the Swiss health care system. J Affect Disord. 2010 May;122(3):224-31. doi: 10.1016/j.jad.2009.07.007. Epub 2009 Aug 8. PMID 19666195
- [Background] Thimm JC, Antonsen L. Effectiveness of cognitive behavioral group therapy for depression in routine practice. BMC Psychiatry. 2014 Oct 21;14:292. doi: 10.1186/s12888-014-0292-x. PMID 25330912
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Demarzo MM, Montero-Marin J, Cuijpers P, Zabaleta-del-Olmo E, Mahtani KR, Vellinga A, Vicens C, Lopez-del-Hoyo Y, Garcia-Campayo J. The Efficacy of Mindfulness-Based Interventions in Primary Care: A Meta-Analytic Review. Ann Fam Med. 2015 Nov;13(6):573-82. doi: 10.1370/afm.1863. PMID 26553897
- [Background] Dimidjian S, Segal ZV. Prospects for a clinical science of mindfulness-based intervention. Am Psychol. 2015 Oct;70(7):593-620. doi: 10.1037/a0039589. PMID 26436311
- [Background] Fernandez E, Salem D, Swift JK, Ramtahal N. Meta-analysis of dropout from cognitive behavioral therapy: Magnitude, timing, and moderators. J Consult Clin Psychol. 2015 Dec;83(6):1108-22. doi: 10.1037/ccp0000044. Epub 2015 Aug 24. PMID 26302248
- [Background] Fjorback LO, Arendt M, Ornbol E, Walach H, Rehfeld E, Schroder A, Fink P. Mindfulness therapy for somatization disorder and functional somatic syndromes: randomized trial with one-year follow-up. J Psychosom Res. 2013 Jan;74(1):31-40. doi: 10.1016/j.jpsychores.2012.09.006. Epub 2012 Oct 1. PMID 23272986
- [Background] Godfrin KA, van Heeringen C. The effects of mindfulness-based cognitive therapy on recurrence of depressive episodes, mental health and quality of life: A randomized controlled study. Behav Res Ther. 2010 Aug;48(8):738-46. doi: 10.1016/j.brat.2010.04.006. Epub 2010 Apr 18. PMID 20462570
- [Background] de Graaf R, Bijl RV, Spijker J, Beekman AT, Vollebergh WA. Temporal sequencing of lifetime mood disorders in relation to comorbid anxiety and substance use disorders--findings from the Netherlands Mental Health Survey and Incidence Study. Soc Psychiatry Psychiatr Epidemiol. 2003 Jan;38(1):1-11. doi: 10.1007/s00127-003-0597-4. PMID 12563553
- [Background] Gu J, Strauss C, Crane C, Barnhofer T, Karl A, Cavanagh K, Kuyken W. Examining the factor structure of the 39-item and 15-item versions of the Five Facet Mindfulness Questionnaire before and after mindfulness-based cognitive therapy for people with recurrent depression. Psychol Assess. 2016 Jul;28(7):791-802. doi: 10.1037/pas0000263. Epub 2016 Apr 14. PMID 27078186
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Hofmeijer-Sevink MK, Batelaan NM, van Megen HJ, Penninx BW, Cath DC, van den Hout MA, van Balkom AJ. Clinical relevance of comorbidity in anxiety disorders: a report from the Netherlands Study of Depression and Anxiety (NESDA). J Affect Disord. 2012 Mar;137(1-3):106-12. doi: 10.1016/j.jad.2011.12.008. Epub 2012 Jan 10. PMID 22240085
- [Background] Jacobi F, Wittchen H-U, Holting C, Hofler M, Pfister H, Muller N, Lieb R. Prevalence, co-morbidity and correlates of mental disorders in the general population: results from the German Health Interview and Examination Survey (GHS). Psychol Med. 2004 May;34(4):597-611. doi: 10.1017/S0033291703001399. PMID 15099415
- [Background] Karsten J, Hartman CA, Smit JH, Zitman FG, Beekman AT, Cuijpers P, van der Does AJ, Ormel J, Nolen WA, Penninx BW. Psychiatric history and subthreshold symptoms as predictors of the occurrence of depressive or anxiety disorder within 2 years. Br J Psychiatry. 2011 Mar;198(3):206-12. doi: 10.1192/bjp.bp.110.080572. PMID 21357879
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kuyken W, Byford S, Taylor RS, Watkins E, Holden E, White K, Barrett B, Byng R, Evans A, Mullan E, Teasdale JD. Mindfulness-based cognitive therapy to prevent relapse in recurrent depression. J Consult Clin Psychol. 2008 Dec;76(6):966-78. doi: 10.1037/a0013786. PMID 19045965
- [Background] Kuyken W, Hayes R, Barrett B, Byng R, Dalgleish T, Kessler D, Lewis G, Watkins E, Morant N, Taylor RS, Byford S. The effectiveness and cost-effectiveness of mindfulness-based cognitive therapy compared with maintenance antidepressant treatment in the prevention of depressive relapse/recurrence: results of a randomised controlled trial (the PREVENT study). Health Technol Assess. 2015 Sep;19(73):1-124. doi: 10.3310/hta19730. PMID 26379122
- [Background] Ma SH, Teasdale JD. Mindfulness-based cognitive therapy for depression: replication and exploration of differential relapse prevention effects. J Consult Clin Psychol. 2004 Feb;72(1):31-40. doi: 10.1037/0022-006X.72.1.31. PMID 14756612
- [Background] Pettersson A, Bostrom KB, Gustavsson P, Ekselius L. Which instruments to support diagnosis of depression have sufficient accuracy? A systematic review. Nord J Psychiatry. 2015;69(7):497-508. doi: 10.3109/08039488.2015.1008568. Epub 2015 Mar 3. PMID 25736983
- [Background] Miller JJ, Fletcher K, Kabat-Zinn J. Three-year follow-up and clinical implications of a mindfulness meditation-based stress reduction intervention in the treatment of anxiety disorders. Gen Hosp Psychiatry. 1995 May;17(3):192-200. doi: 10.1016/0163-8343(95)00025-m. PMID 7649463
- [Background] Pots WT, Meulenbeek PA, Veehof MM, Klungers J, Bohlmeijer ET. The efficacy of mindfulness-based cognitive therapy as a public mental health intervention for adults with mild to moderate depressive symptomatology: a randomized controlled trial. PLoS One. 2014 Oct 15;9(10):e109789. doi: 10.1371/journal.pone.0109789. eCollection 2014. PMID 25333885
- [Background] Roca M, Gili M, Garcia-Garcia M, Salva J, Vives M, Garcia Campayo J, Comas A. Prevalence and comorbidity of common mental disorders in primary care. J Affect Disord. 2009 Dec;119(1-3):52-8. doi: 10.1016/j.jad.2009.03.014. Epub 2009 Apr 10. PMID 19361865
- [Background] Segal ZV, Walsh KM. Mindfulness-based cognitive therapy for residual depressive symptoms and relapse prophylaxis. Curr Opin Psychiatry. 2016 Jan;29(1):7-12. doi: 10.1097/YCO.0000000000000216. PMID 26575299
- [Background] Segal ZV, Bieling P, Young T, MacQueen G, Cooke R, Martin L, Bloch R, Levitan RD. Antidepressant monotherapy vs sequential pharmacotherapy and mindfulness-based cognitive therapy, or placebo, for relapse prophylaxis in recurrent depression. Arch Gen Psychiatry. 2010 Dec;67(12):1256-64. doi: 10.1001/archgenpsychiatry.2010.168. PMID 21135325
- [Background] Stefansson JG, Lindal E. [The prevalence of mental disorders in the Greater-Reykjavik area]. Laeknabladid. 2009 Sep;95(9):559-64. Icelandic. PMID 19738288
- [Background] Stewart-Brown S, Tennant A, Tennant R, Platt S, Parkinson J, Weich S. Internal construct validity of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS): a Rasch analysis using data from the Scottish Health Education Population Survey. Health Qual Life Outcomes. 2009 Feb 19;7:15. doi: 10.1186/1477-7525-7-15. PMID 19228398
- [Background] Strauss C, Cavanagh K, Oliver A, Pettman D. Mindfulness-based interventions for people diagnosed with a current episode of an anxiety or depressive disorder: a meta-analysis of randomised controlled trials. PLoS One. 2014 Apr 24;9(4):e96110. doi: 10.1371/journal.pone.0096110. eCollection 2014. PMID 24763812
- [Background] Sundquist J, Lilja A, Palmer K, Memon AA, Wang X, Johansson LM, Sundquist K. Mindfulness group therapy in primary care patients with depression, anxiety and stress and adjustment disorders: randomised controlled trial. Br J Psychiatry. 2015 Feb;206(2):128-35. doi: 10.1192/bjp.bp.114.150243. Epub 2014 Nov 27. PMID 25431430
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] van Ravesteijn HJ, Suijkerbuijk YB, Langbroek JA, Muskens E, Lucassen PL, van Weel C, Wester F, Speckens AE. Mindfulness-based cognitive therapy (MBCT) for patients with medically unexplained symptoms: process of change. J Psychosom Res. 2014 Jul;77(1):27-33. doi: 10.1016/j.jpsychores.2014.04.010. Epub 2014 May 5. PMID 24913338
- [Background] Vollestad J, Nielsen MB, Nielsen GH. Mindfulness- and acceptance-based interventions for anxiety disorders: a systematic review and meta-analysis. Br J Clin Psychol. 2012 Sep;51(3):239-60. doi: 10.1111/j.2044-8260.2011.02024.x. Epub 2011 Sep 9. PMID 22803933
- [Background] Kuyken W, Byford S, Byng R, Dalgleish T, Lewis G, Taylor R, Watkins ER, Hayes R, Lanham P, Kessler D, Morant N, Evans A. Update to the study protocol for a randomized controlled trial comparing mindfulness-based cognitive therapy with maintenance anti-depressant treatment depressive relapse/recurrence: the PREVENT trial. Trials. 2014 Jun 10;15:217. doi: 10.1186/1745-6215-15-217. PMID 24916319
- [Background] Williams JM, Crane C, Barnhofer T, Brennan K, Duggan DS, Fennell MJ, Hackmann A, Krusche A, Muse K, Von Rohr IR, Shah D, Crane RS, Eames C, Jones M, Radford S, Silverton S, Sun Y, Weatherley-Jones E, Whitaker CJ, Russell D, Russell IT. Mindfulness-based cognitive therapy for preventing relapse in recurrent depression: a randomized dismantling trial. J Consult Clin Psychol. 2014 Apr;82(2):275-86. doi: 10.1037/a0035036. Epub 2013 Dec 2. PMID 24294837
- [Background] Wittchen HU, Jacobi F. Size and burden of mental disorders in Europe--a critical review and appraisal of 27 studies. Eur Neuropsychopharmacol. 2005 Aug;15(4):357-76. doi: 10.1016/j.euroneuro.2005.04.012. PMID 15961293
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] Piet J, Hougaard E. The effect of mindfulness-based cognitive therapy for prevention of relapse in recurrent major depressive disorder: a systematic review and meta-analysis. Clin Psychol Rev. 2011 Aug;31(6):1032-40. doi: 10.1016/j.cpr.2011.05.002. Epub 2011 May 15. PMID 21802618
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Kuyken W, Warren FC, Taylor RS, Whalley B, Crane C, Bondolfi G, Hayes R, Huijbers M, Ma H, Schweizer S, Segal Z, Speckens A, Teasdale JD, Van Heeringen K, Williams M, Byford S, Byng R, Dalgleish T. Efficacy of Mindfulness-Based Cognitive Therapy in Prevention of Depressive Relapse: An Individual Patient Data Meta-analysis From Randomized Trials. JAMA Psychiatry. 2016 Jun 1;73(6):565-74. doi: 10.1001/jamapsychiatry.2016.0076. PMID 27119968
- [Result] Ansseau M, Dierick M, Buntinkx F, Cnockaert P, De Smedt J, Van Den Haute M, Vander Mijnsbrugge D. High prevalence of mental disorders in primary care. J Affect Disord. 2004 Jan;78(1):49-55. doi: 10.1016/s0165-0327(02)00219-7. PMID 14672796